CLINICAL TRIAL: NCT04218435
Title: Impact of Sacubitril/Valsartan on Quality of Life and Mortality of CKD vs Non-CKD in Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Clinision (Other)
Responsible Party: Sponsor
Other Study IDs: PK/IIS/001
Record Dates: First submitted 2019-12-27; First posted 2020-01-06 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2019-10

CONDITIONS: Heart Failure NYHA Class IV; Heart Failure NYHA Class II
Keywords: chronickindeydisease, qualityoflife
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Sacubitril/valsartan is a combination of a neprilysin inhibitor, sacubitril and an angiotensin II receptor blocker, valsartan.
  The recommended starting dose is one 49/51 mg (sacubitril/valsartan) tablet twice-daily. Double the dose of Sacubitril/valsartan after 2 to 4 weeks to the target maintenance dose of 97/103 mg (sacubitril/valsartan) twice-daily, as tolerated by the patient.
  Reduce the starting dose to 24/26 mg (sacubitril/valsartan) twice-daily for:
  * Patients not currently taking an angiotensin-converting enzyme inhibitor (ACEi) or an angiotensin II receptor blocker (ARB) or previously taking a low dose of these agents.
  * Patients with severe renal impairment (CrCl less than 30 ml/min)
  * Patients with moderate hepatic impairment. (Child Pugh B) Double the dose of Sacubitril/valsartan every 2 to 4 weeks to the target maintenance dose of 97/103 mg (sacubitril/valsartan) twice-daily, as tolerated by the patient
  Interventions: Drug: Sacubitril / Valsartan Oral Tablet

INTERVENTIONS:
Drug: Sacubitril / Valsartan Oral Tablet — Sacubitril/Valsartan is indicated to reduce the risk of cardiovascular death and hospitalization for heart failure in patients with chronic heart failure (NYHA Class II-IV) and reduced ejection fraction.
  Sacubitril/Valsartan is usually administered in conjunction with another heart failure therapies, in place of an ACE inhibitor or other ARB.
  Other Names: Sacvin

SUMMARY:
The two primary goals of it's management are preventing further disease progression(mortality,hospitalizations and deterioration of left ventricular function)and alleviating patient suffering

DETAILED DESCRIPTION:
Heart failure (HF) is emerging as an epidemic in 3rd world countries. Despite significant therapeutic advances, patients with chronic heart failure remain at high risk for HF progression and death. The two primary goals of its management are preventing further disease progression(mortality, hospitalizations and deterioration of left ventricular function)and alleviating patient suffering.Sacubitril /valsartan (previously known as LCZ696) is a first-in-class medicine that contains a neprilysin (NEP )inhibitor(sacubitril) and an angiotensin II receptor blocker (valsartan). NEP is an endopeptidase that metabolizes different vasoactive peptides including natriuretic peptides, bradykinin and Ang -II. In consequence, its inhibition increases mainly the levels of both natriuretic peptides (promoting diuresis, natriuresis and vasodilation) and Ang- II whose effects are blocked by the angiotensin receptor blocker, valsartan (reducing vasoconstriction and aldosterone release).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with heart failure (NYHA class II-IV).
2. LV EF(less than or equal to 40%).
3. eGFR (more than 30 ml/min /1.73m2).

Exclusion Criteria:

1. Symptomatic hypotension.
2. eGFR<30 ml/min/1.73m2 .
3. Serum potassium >5.2mmol/L
4. Angioedema

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 130 patients of heart failure with NYHA (II-IV)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Assess the result on the quality of life through Kansas city cardiomyopathy Questionnaire | 1 year
  comparison of the quality of life questionnaire before and after the treatment of sacubitril/ valsartan
Analyze the result on mortality of heart failure patients through Kansas city cardiomyopathy Questionnaire | 1 year
  Improvement in mortality of heart failure patients after taking treatment of sacubitril/ valsartan.

SECONDARY OUTCOMES:
Incidence of acute kidney injury after taking angiotensin receptor neprilysin inhibitor | 1 year
  changes in the baseline of acute kidney injury, electrolyte imbalance and hemodynamic instability before and after taking treatment of sacubitril valsartan

CONTACTS AND LOCATIONS:
Overall Officials: Shahryar Shiekh, Principal Investigator — Doctors hospital and Medical center, Lahore
Locations (1):
- Doctors hospital and medical center, Lahore, Punjab Province, Pakistan